CLINICAL TRIAL: NCT01283100
Title: A Phase 1, Open Label, Single Sequence, Two-Way Drug Interaction Study Evaluating Plasma GSK2248761 and GSK1379572 Pharmacokinetics in Healthy Adult Subjects
Brief Title: A Drug Interaction Study Evaluating Plasma GSK2248761 and GSK1349572 Pharmacokinetics in Healthy Adult Subjects.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: In a Phase II study in HIV-infected patients there were a number of seizures, although exact causality could not be assessed phase 1 activity was terminated.
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 114122
Record Dates: First submitted 2011-01-06; First posted 2011-01-25 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Infection, Human Immunodeficiency Virus I
Keywords: HIV, GSK2248761, GSK1349572, drug interaction, pharmacokinetics
MeSH Terms: conditions — Infections | interventions — dolutegravir; IDX 899

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): GSK1349572 50mg q24h x 7 days
  Interventions: Drug: GSK1349572
- Treatment B (Experimental): GSK2248761 200mg q24h x 7 days
  Interventions: Drug: GSK2248761
- Treatment C (Experimental): GSK1349572 50mg q24h x 7 days + GSK2248761 200mg q24h x 7 days
  Interventions: Drug: GSK1349572; Drug: GSK2248761

INTERVENTIONS:
Drug: GSK1349572 — 50mg once every 24 hours for 7 days
  Arms: Treatment A; Treatment C
Drug: GSK2248761 — 200 mg once every 24 hours for 7 days
  Arms: Treatment B; Treatment C

SUMMARY:
This is a single-center, open-label, three-period, fixed-sequence cross over study in healthy adult subjects. A total of approximately 16 healthy subjects will be enrolled to provide data from 12 evaluable subjects. Subjects will have a screening visit within 30 days prior to the first dose of study drug, three treatment periods, and a follow-up visit 7-14 days after the last dose of study drug. There will be a washout period between Period 1 and Period 2 but no washout between Period 2 and Period 3. Day 1 of Period 3 will be the day after Day 5 of Period 2.

DETAILED DESCRIPTION:
ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, vital signs, laboratory tests, and electrocardiograms (ECGs).
* A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who: Is pre-menopausal with a documented bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries) or hysterectomy, or is post-menopausal defined as 12 months of spontaneous amenorrhea. A follicle stimulating hormone (FSH) level will be performed to confirm a post-menopausal status. For this study, FSH levels > 40 MlU/ml is confirmatory.
* Male subjects must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until the follow-up visit.
* Body weight less than or equal to 50 kg for men and less than or equal to 45 kg for women and body mass index (BMI) within the range 18.5-31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unfit for the study.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* Unwilling to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* History of regular alcohol consumption within 6 months of the study.
* Unwilling to abstain from alcohol for 48 hours prior to the start of dosing until collection of the final pharmacokinetic sample during each treatment period.
* History or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease.

History/evidence of clinically significant pulmonary disease.

* History/evidence of pancreatitis.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy should be excluded.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.

Note: this does not include plasma donation.

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* AST, ALT, alkaline phosphatase and bilirubin greater than or equal to 1.5xULN (isolated bilirubin >1.5x upper limit of normal (ULN) is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Pregnant females as determined by positive serum pregnancy test at screening or prior to dosing.
* Lactating females.
* The subject's systolic blood pressure is outside the range of 90-140 miligrams of mercury (mmHg), or diastolic blood pressure is outside the range of 45-90 mmHg or heart rate is outside the range of 50-100 beats per minute (bpm) for female subjects or 45-100 bpm for male subjects at Screening and predose Day 1.
* Cardiac conduction abnormalities denoted by any of the following on a single 12-lead ECG at screening or predose Day 1 (a single repeat is allowed for eligibility determination).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Plasma GSK1349572 steady state area under the curve (AUC) 0-tau following 50 mg q24h administration with and without GSK2248761 200 mg q24h | 21 days
Plasma GSK1349572 steady state maximum observed concentration (Cmax) following 50 mg q24h administration with and without GSK2248761 200 mg q24h | 21 days
Plasma GSK1349572 steady state Pre-dose trough concentration at the end of the dosing interval (Ctau) following 50 mg q24h administration with and without GSK2248761 200 mg q24h | 21 days
Plasma GSK1349572 steady state predose concentration (C0) following 50 mg q24h administration with and without GSK2248761 200 mg q24h | 21 days
Plasma GSK1349572 steady state minimum concentration (Cmin) following 50 mg q24h administration with and without GSK2248761 200 mg q24h | 21 days
Plasma GSK2248761 steady state steady state AUC 0-tau following 200 mg q24h administration with and without GSK1349572 50 mg q24h | 21 days
Plasma GSK2248761 steady state Cmax following 200 mg q24h administration with and without GSK1349572 50 mg q24h | 21 days
Plasma GSK2248761 steady state Ctau following 200 mg q24h administration with and without GSK1349572 50 mg q24h | 21 days
Plasma GSK2248761 steady state Cmin following 200 mg q24h administration with and without GSK1349572 50 mg q24h | 21 days
Plasma GSK2248761 steady state C0 following 200 mg q24h administration with and without GSK1349572 50 mg q24h | 21 days

SECONDARY OUTCOMES:
Safety and tolerability parameters, including the number of subjects with adverse events | approximately 42 days
Safety and tolerability parameters, including the number of subjects receiving concurrent medications | approximately 42 days
Safety and tolerability parameters, including change from baseline for clinical laboratory safety assessments | approximately 42 days
Safety and tolerability parameters, including change from baseline for electrocardiogram (ECG) assessments | approximately 42 days
Safety and tolerability parameters, including change from baseline for vital sign (blood pressure and heart rate) assessments | approximately 42 days
GSK1349572 PK parameters including time of occurrence of maximum concentration (tmax) following administration of GSK1349572 50 mg q24h with and without co-administration of GSK2248761 200 mg q24h (Day 7 in Period 1, Period 3) | approximately 28 days
GSK1349572 PK parameters including time of occurrence of minimum concentration (Tmin) following administration of GSK1349572 50 mg q24h with and without co-administration of GSK2248761 200 mg q24h (Day 7 in Period 1, Period 3) | 21 days
GSK1349572 PK parameters including apparent clearance following oral dosing (CL/F) of GSK1349572 50 mg q24h with and without co-administration of GSK2248761 200 mg q24h (Day 7 in Period 1, Period 3) | 21 days
GSK1349572 PK parameters including terminal half life (t½) following administration of GSK1349572 50 mg q24h with and without co-administration of GSK2248761 200 mg q24h (Day 7 in Period 1, Period 3) | 21 days
GSK2248761 PK parameters tmax following administration of GSK2248761 200 mg q24h with and without co-administration of GSK1349572 50 mg q24h (Day 7 in Period 2 and Day 7 in Period 3) | 21 days
GSK2248761 PK parameters tmin following administration of GSK2248761 200 mg q24h with and without co-administration of GSK1349572 50 mg q24h (Day 7 in Period 2 and Day 7 in Period 3). | 21 days
GSK2248761 PK parameters CL/F following administration of GSK2248761 200 mg q24h with and without co-administration of GSK1349572 50 mg q24h (Day 7 in Period 2 and Day 7 in Period 3). | 21 days
GSK2248761 PK parameters t½ following administration of GSK2248761 200 mg q24h with and without co-administration of GSK1349572 50 mg q24h (Day 7 in Period 2 and Day 7 in Period 3). | 21 days
GSK1349572 and GSK2248761 Ctau values on Days 4-7 for each Period | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States